CLINICAL TRIAL: NCT02783352
Title: Efficacy of Microfragmented Lipoaspirate Tissue in Arthroscopic Rotator Cuff Repairs: a Randomized Controlled Study
Brief Title: Efficacy of Microfragmented Lipoaspirate Tissue in Arthroscopic Rotator Cuff Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Pietro Randelli, MD, Full Professor, University of Milan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LipoTendon01
Record Dates: First submitted 2016-03-09; First posted 2016-05-26 (Estimated); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Rotator Cuff Tears
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- treatment group (Experimental): arthroscopic rotator cuff repair + injection of autologous micro-fragmented adipose tissue (10 mL)
  Interventions: Procedure: arthroscopic rotator cuff repair; Procedure: autologous micro-fragmented adipose tissue
- control group (Other): arthroscopic rotator cuff repair only
  Interventions: Procedure: arthroscopic rotator cuff repair

INTERVENTIONS:
Procedure: arthroscopic rotator cuff repair — arthroscopic rotator cuff repair
Procedure: autologous micro-fragmented adipose tissue — injection of autologous micro-fragmented adipose tissue (10 mL) after arthroscopic rotator cuff repair, in dry arthroscopy condition
  Arms: treatment group

SUMMARY:
Increasing the success rate of rotator cuff healing remains a tremendous challenge for orthopedic surgeons, which encourage the development of new biological therapies. Among many approaches, activating resident progenitor cells with the Lipogems® product could be an easy, safe, practical and cost-effective new therapeutic strategy for increasing rotator cuff tendon healing.

The primary goal of this study is to evaluate efficacy of infiltration of autologous micro-fragmented adipose tissue in arthroscopic rotator cuff repair, in terms of gain in post-operative Constant score.

DETAILED DESCRIPTION:
Increasing the success rate of rotator cuff healing remains a tremendous challenge for orthopedic surgeons, which encourage the development of new biological therapies. Among many approaches, the possibility of activating resident stem cells in situ, without the need of isolating them from biopsies and successive in vitro culturing, could represent a very promising therapeutic strategy. Along this line, it has been recently demonstrated that a lipoaspirate product, such as the Lipogems® product, contains and produces growth factors that may activate resident stem cells. Recently, it has been discovered that also the human rotator cuff contains a reservoir of progenitor cells, which can be isolated and expanded in vitro.

The primary goal of this study is to evaluate efficacy of infiltration of autologous micro-fragmented adipose tissue in arthroscopic rotator cuff repair, in terms of gain in post-operative Constant score.

Secondary goals are to evaluate efficacy of infiltration of autologous micro-fragmented adipose tissue in arthroscopic rotator cuff repairs, in terms of post-operative pain reduction, gain in post-operative strength in abduction and external rotation; estimate incidence of re-ruptures at 1 and 2 years post-operatively, quantify the amount of fatty degeneration of the supraspinatus at 1 and 2 years post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* 18< Age < 75 years.
* a full-thickness tear of the supraspinatus and/or infraspinatus tendons (classified according to Snyder as degree C1, C2, C3).
* Indication for arthroscopic rotator cuff repair.
* Patients able to understand the study conditions and willing to participate for its entire duration.
* Patients who signed written informed consent.

Exclusion Criteria:

* Patients diagnosed with partial supraspinatus/infraspinatus tears (A1, A2, A3, A4, B1, B2, B3, B4 in Snyder classification system).
* Patients diagnosed with massive rotator cuff tears C4 in Snyder classification system).
* Patients diagnosed with subscapularis tears, of grade III, IV or V in Lafosse classification.
* Patients diagnosed with anterior, posterior or multidirectional shoulder instability.
* Patients diagnosed with Superior Labrum Anterior-to-Posterior (SLAP)-type long-head of the biceps tendon lesions.
* Patients presenting serious comorbidities, which represent contraindications to shoulder arthroscopy.
* Patients treated with hyaluronic acid or steroid intra-articular injections in the index shoulder less than 3 months before the procedure.
* Patients diagnosed with local (shoulder, site of fat tissue harvest or nearby tissues) or systemic infections, osteomyelitis, sepsis.
* Fatty degeneration/atrophy grade III or IV (Goutallier or Fuchs classification) in supraspinatus or infraspinatus muscle bellies.
* Patients diagnosed with diabetes
* Patients diagnosed with chronic kidney disease with Glomerular Filtration Rate (GFR) less than 60 mL/min.
* Patients diagnosed with any disease of coagulation or platelet aggregation systems, or treated with oral anti-coagulating or anti-aggregating agents for which no suspension is possible at the moment of intervention.
* Patients chronically treated with immune-suppressants agents.
* Patients affected by chronic heart failure.
* Patients diagnosed with acute coronary or cerebrovascular disease in the last 6 months.
* Patients who reported weight loss greater than 30 kg for any reasons in the last 12 months or, if the cause is unknown, greater than 10 kg in the last 12 months if the cause
* Patients diagnosed with eating disorders or body dysmorphic disorders.
* Patients with untreated hypo- or hyperthyroidism.
* Patients with varicose veins, phlebitis or scars near the fat tissue harvest area.
* Drug-addicted, alcohol-addicted patients, patients with psychiatric disorders or other clinical conditions, which could compromise the results of the surgical procedure or of the follow-up.
* Informed consent not accepted.
* Pregnant or breastfeeding women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-02; Primary Completion 2020-04-19 (Actual); Study Completion 2021-04-27 (Actual)

PRIMARY OUTCOMES:
Comparison of Constant score between the two groups at 6 months post-operatively | 6 months
  Hypothesis: in the treatment group, Constant score at 6 months post-operatively is at least 7 points HIGHER than Constant score in the control group.

SECONDARY OUTCOMES:
Comparison of Constant score between the two groups at 1, 3, 6, 12, 18, 24 months post-operatively | 1, 3, 6, 12, 18, 24 months
Comparison of ASES score between the two groups at 1, 3, 6, 12, 18, 24 months post-operatively | 1, 3, 6, 12, 18, 24 months
Comparison of Visual Analogue Scale (VAS) difference between the two groups at 1, 3, 7, 14, 30 days and 3, 6, 12, 18, 24 months post-operatively. | 1, 3, 7, 14, 30 days and 3, 6, 12, 18, 24 months
Comparison SST score (simple shoulder test) between the two groups at 1, 3, 6, 12, 18, 24 months post-operatively. | 1, 3, 6, 12, 18, 24 months
Comparison of strength in abduction and external rotation between the two groups at 1, 3, 6, 12, 18, 24 months post-operatively. | 1, 3, 6, 12, 18, 24 months
  Strength will be measured with a dynamometer, using International System metrics.
Comparison of incidence of re-ruptures between the two groups at 18 months post-operatively, measured with magnetic resonance imaging. | 18 months
Comparison of development of fatty degeneration in the supraspinatus at 18 months post-operatively | 18 months
  degeneration is measured with magnetic resonance imaging and classified using the Fuchs classification (grading I-IV)
Number of adverse events for any cause | 7 days, 45-90 days, 12-18 months

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Randelli, MD, Principal Investigator — U.O.C. 1a Divisione, Azienda Socio Sanitaria Territoriale Centro Specialistico Ortopedico Traumatologico Gaetano Pini-CTO
Locations (2):
- Italy (2):
  - U.O.C. 1a Divisione, Azienda Socio Sanitaria Territoriale Centro Specialistico Ortopedico Traumatologico Gaetano Pini-CTO, Milan, Milan
  - IRCCS Policlinico San Donato, San Donato Milanese, Milan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Randelli PS, Cucchi D, Fossati C, Boerci L, Nocerino E, Ambrogi F, Menon A. Arthroscopic Rotator Cuff Repair Augmentation With Autologous Microfragmented Lipoaspirate Tissue Is Safe and Effectively Improves Short-term Clinical and Functional Results: A Prospective Randomized Controlled Trial With 24-Month Follow-up. Am J Sports Med. 2022 Apr;50(5):1344-1357. doi: 10.1177/03635465221083324. Epub 2022 Mar 18. PMID 35302901